CLINICAL TRIAL: NCT05036226
Title: Combination of Autophagy Selective Therapeutics (COAST) in Advanced Solid Tumors or Relapsed Prostate Cancer, A Phase I/II Trial
Brief Title: COAST Therapy in Advanced Solid Tumors and Prostate Cancer
Acronym: COAST
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 103352
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer Recurrent; Solid Tumor, Adult
MeSH Terms: interventions — Hydroxychloroquine; Metformin; Sirolimus; Nelfinavir; Dasatinib

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in sequence of dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose level 1 (Experimental)
  Interventions: Combination Product: Hydroxychloroquine, Metformin, Sirolimus
- Dose level 2a (Experimental)
  Interventions: Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Dasatanib
- Dose level 2b (Experimental)
  Interventions: Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir
- Dose level 3a (Experimental)
  Interventions: Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir, Dasatinib
- Dose level 3b (Experimental)
  Interventions: Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir
- Dose level 4 (Experimental)
  Interventions: Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir, Dasatinib

INTERVENTIONS:
Combination Product: Hydroxychloroquine, Metformin, Sirolimus — Hydroxychloroquine 600mg twice daily Metformin 500mg daily for 7 days, then increase to 1000mg daily Sirolimus 0.5mg daily
  Arms: Dose level 1
Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Dasatanib — Hydroxychloroquine 600mg twice daily Metformin 500mg daily for 7 days, then increase to 1000mg daily Sirolimus 0.5mg daily Dasatinib 20mg daily
  Arms: Dose level 2a
Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir — Hydroxychloroquine 600mg twice daily Metformin 500mg daily for 7 days, then increase to 1000mg daily Sirolimus 0.5mg daily Nelfinavir 1250mg twice daily
  Arms: Dose level 2b
Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir, Dasatinib — Hydroxychloroquine 600mg twice daily Metformin 500mg daily for 7 days, then increase to 1000mg daily Sirolimus 0.5mg daily Nelfinavir 1250mg twice daily Dasatanib 20mg daily
  Arms: Dose level 3a
Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir — Hydroxychloroquine 600mg twice daily Metformin 500mg daily for 7 days, then increase to 1000mg daily Sirolimus 0.5mg daily Nelfinavir 2500mg twice daily
  Arms: Dose level 3b
Combination Product: Hydroxychloroquine, Metformin, Sirolimus, Nelfinavir, Dasatinib — Hydroxychloroquine 600mg twice daily Metformin 500mg daily for 7 days, then increase to 1000mg daily Sirolimus 0.5mg daily Nelfinavir 2500mg twice daily Dasatanib 20mg daily
  Arms: Dose level 4

SUMMARY:
The purpose of this Phase I/II study is to determine the safety and effectiveness of up to 5 study drugs used together for the treatment of solid tumor cancers. The drugs are hydroxychloroquine, metformin, sirolimus, dasatinib and nelfinavir and are given orally.

DETAILED DESCRIPTION:
This is a Phase I/II safety and efficacy study of COAST therapy in patients with advanced cancer for which no satisfactory therapy options exist. An initial Phase I cohort of 18-30 patients with advanced cancer will receive increasing components of the COAST regimen following a traditional 3+3 escalation design. The starting COAST combination includes hydroxychloroquine, sirolimus and metformin (DL1 - base combination). If this three-drug base combination is cleared for safety, two dose levels will be opened for enrollment exploring the safety of the base in combination with either dasatinib or nelfinavir. Patients will be assigned sequentially to DL2A (base + dasatinib) and DL2B (base + nelfinavir). If nelfinavir is deemed unsafe in combination with the base (DL2B is not cleared for safety, regardless of the safety of DL2A), no further drug combinations will be explored since all remaining combinations include nelfinavir. If both dasatinib and nelfinavir are individually safe in combination with the base (DL2A and DL2B are both cleared for safety), two additional dose levels will be explored, the first combining all five drugs and the second exploring nelfinavir at a higher dose. If dasatinib is not safe but nelfinavir is safe in combination with the base (DL2A but not DL2B cleared for safety), then only one additional dose level will be explored combining the base with a higher dose of nelfinavir. If neither DL2A nor DL2B are cleared for safety, then only the base combination may be considered safe. Once a given dose level is cleared for initial DLT evaluation (e.g., 0 of 3 patients have a DLT or at most 1 of 6 have a DLT), additional patients may be enrolled (i.e., 'backfilled') to that dose level while a higher dose level is being evaluated for safety. Prioritization for backfill will be given to dose levels proximal to the current dose level being explored, and to those dose levels with evidence of anti-tumor activity. Backfill patients who are DLT-evaluable will be included in making decisions on dose escalation. Accrual to a dose-level may be halted and additional patients enrolled to a lower dose level that was previously cleared for safety depending on the total number of DLTs observed among all DLT-evaluable patients at that lower dose level (initial and backfill patients). The maximum tolerated mixture is the highest dose level at which at most 1 of 6 patients experiences a DLT or, for a dose level sample size >6 due to additional backfill patients, the highest dose level at which the observed DLT rate is ≤16.7%. The recommended phase 2 dose (RP2D) will be determined based on the totality of data, including the maximum tolerated mixture, dose adjustments, all safety data including any DLT-equivalent events (safety events that meet the criteria for a DLT regardless of treatment cycle and trial phase), and any response data. The study team may recommend a dose level lower than the maximum tolerated mixture as the RP2D based on their review of the data in aggregate. However, the RP2D will not exceed the dose level corresponding to the maximum tolerated mixture. The phase II efficacy trial will evaluate the anti-tumor activity of the COAST RP2D combination in patients with advanced prostate cancer based on a Simon two stage optimum design. The primary endpoint is the16-week PSA progression-free rate following treatment initiation, where PSA progression is defined per PCWG3. A maximum of 29 patients will be enrolled. In the first stage, 10 patients will be accrued. If none of the first 10 patients are PSA progression-free at 16 weeks, we will halt registration. If one or more patients are PSA progression-free at 16 weeks, an additional 19 patients will be enrolled. If 4 or more out of the 29 patients are PSA progression-free at 16 weeks, the treatment will be declared promising. This study is powered at 80% with a one-sided type I error rate of 5%. Specifically, this study has an 80% chance of declaring promise if the true 16-week PSA progression-free rate is at least 20%. If instead the true 16-week PSA progression-free rate is at most 5%, then the study has a 5% chance of declaring promise and a 60% chance of early termination. Phase I patients treated at the RP2D who meet inclusion and exclusion criteria for phase II will be included in the phase II cohort. Treatment will continue until there is 1) unacceptable toxicity (grade 3 or 4 toxicity that does not resolve to grade 1 or less by 28 days after drug withdrawal), 2) institution of new additional cancer therapy, 3) withdrawal of consent, 4) any condition that, in the opinion of the treating physician, renders continued COAST treatment to not be in the patient's best interest, 5) lack of compliance with study procedures by the patient, or 6) PSA progression by 16 weeks of COAST therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have advanced solid tumor cancer of any type (Phase I) or advanced prostate cancer (Phase II). Prostate cancer patients must have a PSA of at least 0.1 ng/mL.
2. Tissue diagnosis documented by pathology report, or clinic note attesting to same.
3. Measurable / evaluable tumor by RECIST, quantitative blood biomarker, or radionuclide imaging
4. Voluntary, signed and dated, Institutional Review Board (IRB) approved consent form in accordance with regulatory and institutional guidelines.
5. Documented progression of disease during treatment with one or more standard systemic regimens. Single or multiple regimens of chemotherapy, hormone suppression therapy, radiation therapy, surgery, immunotherapy, or adoptive cell therapy are allowed.
6. 18 years of age or older.
7. ECOG performance status of 0-2.
8. Bilirubin ≤ 1.5 times upper limit of normal (ULN) and AST / ALT ≤ 3 times ULN. Subjects with Gilbert's syndrome may be included if the total bilirubin is < 3 times ULN and the direct bilirubin is within normal limits.
9. Serum creatinine ≤ 1.5 times ULN.
10. Absolute neutrophil count (ANC) ≥ 1,000 cells / mm3
11. Platelet count ≥ 75,000 cells / mm3
12. Hemoglobin ≥ 9 g/ dL.
13. Fasting glucose ≤ 160 mg/dL or non-fasting glucose ≤ 200 mg/dL.
14. Urinalysis with no clinically significant abnormalities.
15. Adequately controlled blood pressure as determined by the treating investigator.
16. Subjects with the potential to produce children must agree to effective contraceptive method use during study participation.
17. Patients requiring narcotic analgesics must be on stable doses for at least 2 weeks prior to study entry.
18. Patients being considered for a dose level containing nelfinavir mesylate must discontinue any statin use within 48 hours of beginning study treatment.

Exclusion Criteria:

1. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or history of ischemia on ECG.
2. Underlying psychiatric disorder requiring hospitalization within the last two years.
3. Clinically significant neurological disorder (Parkinson's disease, dementia, multiple sclerosis), as determined by the enrolling investigator.
4. Active, uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy.
5. Treatment with local or systemic radiation therapy, surgery, or investigational therapy within 28 days prior to registration.
6. Unwillingness or inability to comply with procedures required in this protocol.
7. Serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator.
8. Patients who are receiving, coumadin, apixaban, argatroban or rivaroxaban.
9. Patients who are currently participating in any other clinical trial of an investigational product.
10. Any other mental incapacitation or psychiatric illness that would preclude study participation, as determined by the enrolling investigator.
11. Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) - Phase I | Minimum of 3 months after start of treatment on each dose level
  Maximum dose achievable without dose limiting toxicities (DLT's)
Measure of proportion of patients with disease control - Phase II | Minimum of 16 weeks after start of treatment, per patient
  Stable disease by RECIST or PCWG3 criteria after 16 weeks of treatment on study.

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) score | Minimum of 16 weeks of treatment on study
  To document the change in QOL (via disease-specific FACT questionnaire, composite score) in patients treated with COAST) after two and four cycles of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States